CLINICAL TRIAL: NCT05374993
Title: An Early Feasibility Evaluation of a Novel 3rdMolarTooth Bud Ablation Procedure
Acronym: 3TBA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding limitation
Sponsor: TriAgenics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TP-015
Record Dates: First submitted 2022-05-06; First posted 2022-05-16 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Molar, Third

STUDY DESIGN:
Intervention Model Description: Single-arm prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 3TBA Procedure (Experimental)
  Interventions: Device: 3TBA

INTERVENTIONS:
Device: 3TBA — Induce third molar tooth bud agenesis

SUMMARY:
This single-arm prospective study will enroll a minimum of 7 and a maximum 10 subjects between the ages of 7 and 13 years of age with radiographic evidence of mandibular 3rd molar tooth bud development without enamel formation. Each subject will undergo a 3TBA procedure for each qualifying mandibular 3rd molar tooth buds. Each subject will receive treatment for qualifying mandibular tooth buds during the same session. Subjects will be followed for a minimum of 12 weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 7 and 13 years of age
2. Subject has radiographic evidence of at least one mandibular 3rd molar tooth bud

Exclusion Criteria:

1. Subject use of articaine is contraindicated (known hypersensitive to products containing sulfites).
2. Subject has any condition which, in the opinion of the Investigator, would prevent adequate performance of the procedure or affect the health and/or safety of the subject.-

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Tooth Structure Development Assessment | 12 weeks
  Efficacy assessment will be performed based on periapical X-rays from Follow-up Visit 3 (12-week post treatment). Effectiveness Assessment will consist of evaluation of Tooth Structure Development and Bony Crypt In Growth using the following scale.
  Tooth Structure Development Assessment Scale for 3rd Molar:
  "0" = No radiographic evidence.
  "1" = Minimal or trace level of detectable radiographic evidence.
  "2" = Moderate or intermediate level of detectable radiographic evidence of mineralized tooth structure formation with crown formation to be less than 50% complete.
  "3" = Advanced level of detectable radiographic evidence of mineralized tooth structure formation with enamel formation estimated to be 50% or more complete.
  Success is defined as a score of "0" or "1" on Tooth Structure Development scale at Follow-up Visit 3 (12-week post treatment). Each treated tooth bud is evaluated individually.
Bony Crypt Growth Assessment | 12 weeks
  Efficacy assessment will be performed based on periapical X-rays from Follow-up Visit 3 (12-week post treatment). Effectiveness Assessment will consist of evaluation of Bony Crypt In Growth using the following scales.
  Tooth Structure Development Assessment Scale for 3rd Molar:
  "0" = No radiographic evidence.
  "1" = Minimal or trace level of detectable radiographic evidence of mineralized tooth structure formation.
  "2" = Moderate or intermediate level of detectable radiographic evidence of mineralized tooth structure formation with crown formation to be less than 50% complete.
  "3" = Advanced level of detectable radiographic evidence of mineralized tooth structure formation with enamel formation estimated to be 50% or more complete.
  N/I = Not Interpretable. N/A = Not Applicable.
  Success is defined as a score of "0" or "1" on Bony Crypt Growth Assessment scales at Follow-up Visit 3 (12-week post treatment). Each treated tooth bud is evaluated individually.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12 weeks
  * Proximal second molars continue to erupt normally
  * Proximal second molars have no radiographic evidence of crown alteration
  * Surgical site is completely healed over on visual exam
  * Radiographic assessment of the surgical site is WNL expected or post op healing
  * No adverse events related to the 3TBA procedure
  * No reported neurological changes to tongue or lip

IPD SHARING:
Plan to Share IPD: No